CLINICAL TRIAL: NCT04449549
Title: Rapid Analysis and Response Evaluation of Combination Anti-Neoplastic Agents in Rare Tumors (RARE CANCER) Trial: RARE 1 Nilotinib and Paclitaxel
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200121; 20-C-0121
Record Dates: First submitted 2020-06-26; First posted 2020-06-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11-28

CONDITIONS: Neoplasms
Keywords: Pharmacodynamic; BCR Abl kinase inhibitor; Taxanes; Combination
MeSH Terms: conditions — Neoplasms | interventions — nilotinib; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Nilotinib will be administered at 300 mg orally BID; Paclitaxel will be administered IV at 80 mg/m2 on Days 1, 8, and 15 in 28-day cycles.
  Interventions: Drug: Nilotinib and Paclitaxel

INTERVENTIONS:
Drug: Nilotinib and Paclitaxel — The BCR-Abl kinase inhibitor nilotinib demonstrated greater than additive activity in combination with the anti-tubulin agent paclitaxel in preclinical xenograft models, justifying the clinical evaluation of this combination for its antitumor activity

SUMMARY:
Background:

People with rare cancers often have limited treatment options. The biology of rare cancers is not well understood. Researchers want to find better treatments for these cancers. They want to test 2 drugs that, taken separately, have helped people with non-rare cancers. They want to see if these drugs together can make rare cancers shrink or stop growing.

Objective:

To learn if nilotinib and paclitaxel will benefit people with rare cancers.

Eligibility:

People age 18 and older who have a rare, advanced cancer that has progressed after receiving standard treatment, or for which no effective therapy exists.

Design:

Participants will be screened with medical history and physical exam. They will have blood and urine tests. They will have a pregnancy test if needed. They will have an electrocardiogram to check their heart. They will have imaging scans to measure their tumors.

Participants will repeat the screening tests during the study.

Participants will receive nilotinib and paclitaxel. The drugs are given in 28-day cycles. Nilotinib is a capsule taken by mouth twice a day. Paclitaxel will be given intravenously by peripheral line or central line once a week for the first 3 weeks of each cycle.

Participants will keep a medicine diary. They will track when they take the study drugs and any side effects they may have.

Participants may have optional tumor biopsies.

Participants can stay on the study until their disease gets worse or they have intolerable side effects.

Participants will have a follow-up phone call about 30 days after taking the last dose of study drugs....

DETAILED DESCRIPTION:
Background:

* Rare tumors constitute a heterogeneous group of cancers associated with limited treatment options and poor outcomes. Due to their rarity, there are few good models for these diseases to support preclinical evaluation of new anticancer agents. To address these challenges, DCTD s Patient-Derived Models Repository (PDMR) is generating patient-derived xenograft models of adult and pediatric rare cancers and has screened combinations of approved and investigational anticancer agents in these models.
* Based on preclinical activity, drug combinations are being tested in patients with rare cancers in a series of connected Phase 2 clinical trials (Rapid Analysis and Response Evaluation of Combination Anti-Neoplastic Agents in Rare Tumors [RARE CANCER]); responses may trigger further evaluation of a treatment in that rare cancer type to further evaluate response rate and mechanism-of-action. Patients who progress will be offered another RARE CANCER trial.
* The agents used in this trial are the BCR-Abl kinase inhibitor nilotinib and the anti-tubulin agent paclitaxel, which showed greater than additive activity in combination in preclinical xenograft models and subsequently demonstrated clinical efficacy (including partial responses) in patients with solid tumors on the Phase 1 trial 15-C-0086 (NCT02379416).

Primary Objectives:

- To evaluate the proportion of patients with advanced rare cancers who have objective responses (OR) to treatment with nilotinib and paclitaxel

Exploratory Objectives:

* To evaluate the proportion of patients alive and progression free at 6 months on study agents
* To identify genomic and transcriptomic determinants of response and resistance in tumor biopsy specimens
* To examine genomic alterations in circulating tumor DNA (ctDNA) and circulating tumor cells (CTCs) that may be associated with response or resistance
* To evaluate the pharmacodynamic effects of the combination on biomarkers of cell death and epithelial-to-mesenchymal transition in tumor tissue and CTCs

Eligibility:

* Study participants must have a histologically confirmed solid tumor meeting the RARECARE definition of rare tumor that has progressed on standard therapy known to prolong survival or for which no standard treatment options exist; with Mod G (6-17-24), eligibility will be limited to patients with granulosa cell ovarian cancer, clear cell ovarian cancer, anal cancer, or Ewing sarcoma.
* Age >= 18
* No major surgery, radiation, or chemotherapy within 3 weeks prior to entering the study (6 weeks for nitrosoureas and mitomycin C) or 5 half-lives of the agent, whichever is shorter; toxicity from prior treatment must have recovered to eligibility levels.
* Adequate organ function; performance status ECOG 0-2

Study Design:

* Nilotinib will be administered at 300 mg orally BID and paclitaxel will be administered IV at 80 mg/m^2 on Days 1, 8, and 15 in 28-day cycles.
* A single-stage design will be used with a target accrual of 30 eligible patients. If at least 4/30 patients experience an objective response (PR or CR by RECIST 1.1), the combination of nilotinib and paclitaxel will be considered promising. The accrual ceiling is 34 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed rare solid tumors that have progressed on standard therapy known to prolong survival or for which no standard treatment options exist. The list of eligible rare tumors can be found below**. With Amendment G (v 6-17-24), eligibility will be limited to patients with adult granulosa cell ovarian cancer, clear cell ovarian cancer, anal cancer, or Ewing sarcoma.Patients must have measurable and evaluable disease.
* Age >= 18 years.
* ECOG performance status <= 2.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count >=1,500/mcL
  * Platelets >=100,000/mcL
  * Total bilirubin <=1.5 X institutional ULN
  * AST(SGOT)/ALT(SGPT) <=3 X institutional upper limit of normal; <= 5.0 x ULN in patients with liver metastases
  * creatinine <=1.5 X institutional ULN OR
  * creatinine clearance >=60 mL/min/1.73 m^2 for patients with creatinine levels >1.5 mg/dL
* Nilotinib and paclitaxel have both been assigned to pregnancy category D by the FDA. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for at least 3 months after dosing with study drugs ceases. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of study drug administration.
* Patients must have completed radiation therapy or major surgery >= 3 weeks, or biologic therapy or chemotherapy >= 5 half-lives or 3 weeks, whichever is shorter (6 weeks for nitrosoureas and mitomycin C) prior to entering the study. Patients must be >= 2 weeks since any prior administration of a study drug in a Phase 0 or equivalent study and be >= 1 week from palliative radiation therapy (patients on study may be eligible for palliative radiotherapy to non-targeted lesions after 2 cycles of therapy at the PI s discretion). Patients must have recovered to eligibility levels from prior toxicity or adverse events. Treatment with bisphosphonates is permitted.
* Biopsies are optional on this study. In lieu of baseline biopsies, patients are encouraged to submit at registration archival tumor biopsy tissue from a previous research study or medical care providing it meets the minimum collection and preservations requirements outlined for the submission of archival tissue are:

  * Tissue must have been collected within 3 months prior to registration.
  * Patient must not have received any intervening therapy for their cancer since the collection of the tumor sample.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. For these patients, an HIV viral load test must be completed within 28 days prior to enrollment.

  * Rare Tumor Eligibility List

    1. Epithelial tumors of nasal cavity, sinuses, nasopharynx
    2. Epithelial tumors of major salivary glands
    3. Salivary gland type tumors of head and neck, lip, esophagus, stomach, trachea and lung, breast and other location
    4. Undifferentiated carcinoma of gastrointestinal (GI) tract
    5. Adenocarcinoma with variants of small intestine
    6. Squamous cell carcinoma with variants of GI tract (stomach small intestine, colon, rectum, pancreas)
    7. Fibromixoma and low-grade mucinous adenocarcinoma (pseudomixoma peritonei) of the appendix and ovary
    8. Rare Pancreatic tumors including acinar cell carcinoma, mucinous cystadenocarcinoma or serous cystadenocarcinoma
    9. Intrahepatic cholangiocarcinoma
    10. Extrahepatic cholangiocarcinoma and bile duct tumors
    11. Sarcomatoid carcinoma of lung
    12. Bronchoalveolar carcinoma lung (a.k.a. adenocarcinoma in situ, minimally invasive adenocarcinoma, lepidic predominant adenocarcinoma, or invasive mucinous adenocarcinoma)
    13. Non-epithelial tumors of the ovary
    14. Trophoblastic tumor
    15. Transitional cell carcinoma other than that of the renal, pelvis, ureter, or bladder
    16. Cell tumor of the testes and extragonadal germ tumors
    17. Epithelial tumors of penis - squamous adenocarcinoma cell carcinoma with variants of penis
    18. Squamous cell carcinoma variants of the genitourinary (GU) system
    19. Spindle cell carcinoma of kidney, pelvis, ureter
    20. Adenocarcinoma with variants of GU system (excluding prostate cancer)
    21. Odontogenic malignant tumors
    22. Pancreatic neuroendocrine tumor (PNET)
    23. Neuroendocrine carcinoma including carcinoid of the lung
    24. Pheochromocytoma, malignant
    25. Paraganglioma
    26. Carcinomas of pituitary gland, thyroid gland parathyroid gland and adrenal cortex
    27. Desmoid tumors
    28. Peripheral nerve sheath tumors and NF1-related tumors
    29. Malignant giant cell tumors
    30. Chordoma
    31. Adrenal cortical tumors
    32. Tumor of unknown primary (Cancer of Unknown Primary; CuP)
    33. Not Otherwise Categorized (NOC) Rare Tumors
    34. Adenoid cystic carcinoma
    35. Vulvar cancer
    36. MetaPLASTIC carcinoma (of the breast)
    37. Gastrointestinal stromal tumor (GIST)
    38. Perivascular epithelioid cell tumor (PEComa)
    39. Apocrine tumors/Extramammary Paget s Disease
    40. Peritoneal mesothelioma
    41. Basal cell carcinoma
    42. Clear cell cervical cancer
    43. Esthenioneuroblastoma
    44. Endometrial carcinosarcoma (malignant mixed Mullerian tumors)
    45. Clear cell endometrial cancer
    46. Clear cell ovarian cancer
    47. Gestational trophoblastic disease (GTD)
    48. Gallbladder cancer
    49. Small cell carcinoma of the ovary, hypercalcemic type
    50. Angiosarcoma
    51. High-grade neuroendocrine carcinoma
    52. Treatment-emergent small-cell neuroendocrine prostate cancer (t-SCNC)
    53. Anal cancer
    54. Lymphoma
    55. Merkel cell carcinoma
    56. Pleural Mesothelioma
    57. Sarcoma (bone & soft tissue)
    58. Thymic Carcinoma
    59. Uterine Leiomyosarcoma
    60. Papillary RCC

EXCLUSION CRITERIA:

* QTcF interval of >=450 msec at study entry; congenital long QT syndrome
* Sensory/motor neuropathy >= Grade 2
* Patients who are receiving any other investigational agents.
* Patients with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases are excluded, with the following exceptions:

  * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, or cerebellum
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted.
    * No neurosurgical resection or brain biopsy within 28 days prior to Cycle 1, Day 1
  * Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

    * Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and radiographic screening for the current study
    * No stereotactic radiation or whole-brain radiation within 28 days prior to Cycle 1, Day 1
    * Screening CNS radiographic study >=4 weeks from completion of radiotherapy and >=2 weeks from discontinuation of corticosteroids
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs.
* Uncontrolled intercurrent illness including, but not limited to, serious untreated infection, symptomatic respiratory failure/congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because nilotinib and paclitaxel have been assigned to pregnancy category D by the FDA. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued prior to the first dose of study drug and women should refrain from nursing throughout the treatment period and for 3 months following the last dose of study drug.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Objective response | 12 months
  If at least 4/30 patients experience an objective response, defined as a complete or partial response by RECIST 1.1, the combination of nilotinib and paclitaxel will be considered promising. This design provides approximately 88% power to reject a null ORR of 0.05 when the true ORR is 0.2 (with one-sided type-I error of approximately 0.062).

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kummar S, Chen HX, Wright J, Holbeck S, Millin MD, Tomaszewski J, Zweibel J, Collins J, Doroshow JH. Utilizing targeted cancer therapeutic agents in combination: novel approaches and urgent requirements. Nat Rev Drug Discov. 2010 Nov;9(11):843-56. doi: 10.1038/nrd3216. Epub 2010 Oct 29. PMID 21031001
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0121.html